| A Randomized Factorial Feasibility Study of High-Resistance Circuit Training | |
|---|---|
| Strength Training Intervention in Untrained Adolescents: A Mixed Metho | ods Approach |

Mitchell Wyatt<sup>1</sup>, Leslie Podlog<sup>2</sup>, Ryan Burns<sup>1</sup>, Bradley King<sup>1</sup>, Kristin Heumann<sup>3</sup>, and Timothy Brusseau Jr.<sup>1</sup>

**NCT: TBA** 

11/20/24

Correspondence:

Mitchell Wyatt

mitch.wyatt@utah.edu

Quebec.

<sup>&</sup>lt;sup>1</sup>Department of Health and Kinesiology, University of Utah, Salt Lake, Utah.

<sup>&</sup>lt;sup>2</sup>School of Kinesiology and Physical Activity Sciences, University of Montreal, Montreal,

<sup>&</sup>lt;sup>3</sup>Department of Kinesiology, Colorado Mesa University, Grand Junction, Colorado.

#### Methods

# **Experimental design**

This study used an explanatory sequential design by collecting quantitative data first, then qualitative data to expand understanding of participant experience. After receiving University of Utah IRB and Murray School District Board approval, a cohort of participants were recruited for a before-school trial. Due to low enrollment of the before-school trial, another cohort of participants were recruited for an after-school trial following the conclusion of the before-school trial. Before-school sessions were conducted October 23<sup>rd</sup> to November 17<sup>th</sup> at 6:30 AM to 7:50 AM. After-school sessions were conducted November 27th to December 14th at 2:40 PM to 4:00 PM. After obtaining parental consent and participant assent, participants completed a pre-intervention testing session. Using randomizing software from randomizer.org, participants were randomized and stratified by sex into the high-resistance circuit training group (HRC) or traditional strength training group (ST). A waitlist control group was part of the original experimental design, however due the small sample, it was removed. The training section below contains details on the training protocols for the different groups. Concluding the intervention, subjects completed post-intervention testing. Primary feasibility outcomes included: consent rate, fidelity, participant attendance, study retention, adverse events, and participant experience. Secondary outcomes included measures of strength, body composition and aerobic fitness. After the conclusion of the intervention and quantitative data analysis, participants were invited for a one month follow up interview assessing their motivation to join the study, barriers and experiences partaking in the study.

## **Participants**

Seven healthy untrained adolescents (16.9 ± .7 years old, 4 males and 3 females) from a northern Utah high school participated. The high school had 1,500 students across 10<sup>th</sup>, 11<sup>th</sup> and 12<sup>th</sup> grades. For the purpose of this study, untrained participants were defined as participants who reported being physically inactive with no regular participation in physical activity for the past month prior to the intervention. Participants were recruited through posted flyers and table events during lunch periods. Exclusion criteria included recent injuries or medical conditions that may influence high-intensity performance, currently enrolled in another training program including resistance, cardiovascular, or sports-based program, uninsured participants, drastically altering diet and use of performance-enhancing substances (i.e., creatine, pre-workout, post-workout supplements). Prior to the start of the study, participants and respective guardians read and signed informed consent, parent permission and assent documents. The 2023 PAR-Q + form and modified Copper Institute Fitnessgram and Activitygram questionnaires were used to screen participants.

**Table 1. Summary Table of Participants** 

| Category | Frequency | Percent |
|--------------|-----------|----------|
| Sex | | <u> </u> |
| Male | 4 | 57% |
| Female | 3 | 43% |
| Ethnicity | I | <u>l</u> |
| Non-Hispanic | 7 | 100% |
| Race | | <u> </u> |
| White | 7 | 100% |
| | I | <u>l</u> |

| Category | Mean | Standard Deviation |
|---------------------|------|--------------------|
| Age | 16.9 | 0.7 |
| BMI | 24.4 | 5.8 |
| Body Fat Percentage | 25.3 | 8.9 |

Table 1 shows the baseline participant characteristics.

# Protocol

Participants performed 1-1 ½ hour sessions three times a week for four weeks under the supervision of the primary researcher. Participants followed the weekly progression adapted from Alcarez [32]. Exercises were adapted to fit the facility's equipment by prioritizing free weight compound movements over single joint machine exercises. In addition, instead of prescribing 6RM (85% of 1RM) to untrained participants, an autoregulatory approach using rate of perceived exertion (RPE) was prescribed (Figure 2). To simplify RPE use, participants used whole numbers such as 8 RPE which lowers the intensity from HRC's traditional intensity of 85% of 1RM to 80% 1RM. Literature supports the use of RPE-based loading as an effective alternative to prescribing percentages of 1RM for improving strength [39]. Use of RPE-based loading negated a safety concern with untrained participants conducting 1RM testing.

Figure 2. Equivalent Intensity Prescriptions of Traditional Percentage Based and RPE

| Targeted strength quality | Percent of 1RM | Rate of perceived exertion | Reps left in reserve |
|---|---|---|---|
| Maximal strength | 85% | 8.5 | 1-2 |
| Strength-speed | 80% | 8 | 2 |

Figure 2 shows the equivalent values for percent of 1RM loading vs RPE-based loading adapted from Shattock & Tee [40].

The following four-week progression was developed to help participants become familiar with basic weightlifting movements in addition to appropriately increase intensity of sessions (Figure 3). In the first week of the intervention, ST and HRC groups completed 4 sets of each exercise at 6 RPE on the 1-10 modified Borg Scale. During this time, emphasis was given to proper weightlifting technique over the amount of weight being used. In the second week, participants completed 2 sets of 6 RPE, then 2 sets of 7 RPE. In the third week, participants increased intensity to 2 sets of 7 RPE and 2 sets of 8 RPE. In the fourth week, participants increased intensity to 4 sets of 8 RPE. Participants were expected to complete the workouts and appropriately increase the difficulty of resistance used if movements were performed correctly. Lifts were performed at a tempo with a 3 second eccentric phase, 2 second isometric pause, followed by a concentric phase at maximum velocity. Participants were able to adjust resistance by 2-5% each set based on RPE.

Figure 3. Periodization of Training Volume

| Week 1 | Week 2 | Week 3 | Week 4 |
|-----------------|-----------------|-----------------|-----------------|
| | 2 sets at 6 RPE | 2 sets at 7 RPE | |
| 4 sets at 6 RPE | 2 sets of 7 RPE | 2 sets of 8 RPE | 4 sets at 8 RPE |

Figure 3 shows the progression of prescribed sets across weeks.

# **Training**

Warm Up. Participants in ST and HRC groups engaged in a 5 min warm-up specific to the first block followed by 5 min of dynamic stretching and mobility. Participants then performed 2 sets of the first three exercises using the following sequence; 10 reps at 5 RPE with 30 sec - 1 min rest, 8 reps at 6-7 RPE with 30 sec - 1 min rest, then participants started target sets of 6 reps at the prescribed RPE.

Strength Training. Once the warm-up was completed, ST participants performed the 6 reps of the first exercise at the prescribed RPE then rested 1 minute. Participants then completed another set of their first exercise with the required rest until the prescribed sets were completed. Participants performed the second and third exercise in the same fashion. Once the first block was completed, participants rested 5 min, then completed the second block with the same warm up sequence.

High-Resistance Circuit Training. An adapted version of Alcaraz's HRC was utilized in the intervention. Exercises and intensities used by ST was the same for HRC except HRC participants performed the first three exercises as a circuit with 35 seconds rest between exercises (Figure 4).

Figure 4. Protocols for the ST and HRC Training Groups



Figure 4 shows the Traditional Strength Training (ST) and High-Resistance Circuit Training (HRC) interventions at week 4 of the intervention. ST participants performed four sets of six reps of a single exercise with 1 minute rest between sets. HRC performed the same exercises in a circuit fashion rotating from one exercise to another with 35 sec rest between sets.

## **Feasibility outcomes**

Primary feasibility outcomes included recruitment process, sample size, consent rate, retention rate, fidelity, attendance, participant experience, and adverse events.

Recruitment process. The recruitment process refers to the protocols used to find, select, and enroll participants into a study [41]. The recruitment process for this study was represented by reporting the total number of unique QR code scans from posted flyers and tabling events, the number of completed interest forms, the number of eligible participants and the number of consented participants. A recruitment period of 3 weeks was given for the before and afterschool trials.

Sample size. Sample size was used as another key feasibility marker and refers to the total number of individuals used in the intervention. A sample size of 30 participants per trial with 15 participants in each treatment group was established based on previous literature examining the difference between resistance training groups [32], suggestions of 12 participants minimum per group in feasibility trials from Julious [42], and practicality how many participants could receive intervention treatment with proper supervision. While larger sample sizes would be ideal for secondary fitness outcomes, the primary purpose of this study was to assess feasibility outcomes and not report statically powered differences.

Consent rate. Consent rate is often referred to as the percentage of participants enrolled divided by the number of eligible participants [43]. For this study, consent rate was calculated by taking the total number of participants that consented and were randomized divided by the number of eligible students. An acceptable consent rate was set at 80% based on findings from Jacques [43].

Retention rate. Retention rate is defined as the percentage of the total number of randomized participants assessed for primary outcomes and used in the primary outcome analysis [43]. For the purpose of this study, researchers were interested in retention for both primary and secondary outcomes meaning researchers tracked retention from pre-intervention fitness testing, through treatments, and post-intervention fitness testing sessions. The follow up interview was not included in calculating the retention rate. Only participants that withdrew from the study or were not included in the primary and secondary outcome analysis influenced the retention rate. Thus, retention was calculated as the percentage of participants that completed pre and post-intervention fitness assessments and intervention treatment divided by the number of participants randomized into treatment groups. Participants that withdrew (i.e., stopped attending) from the study were tracked by the investigator. Based on prior literature, 80% retention rate was used as an acceptable threshold [44].

Fidelity. Fidelity is referred to how well an intervention was delivered as intended and is measured at the participant, deliverer or setting level [41]. For this study, fidelity was assessed at the instructor (deliverer) and participant level. Instructor fidelity was measured as a percentage by totaling the provided sessions divided by the total number of planned sessions. An acceptable percentage was set at 80% due to conflicts with events such as holiday breaks or parent teacher conferences. To assess participant fidelity, the primary researcher and participants recorded session durations, completed sets and intensity along with activity and diet audits at weeks 2, and 4 of the intervention. The activity and diet audit included a modified Copper Institute

Fitnessgram and Activitygram questionnaire (Figure 5). If participants recorded additional days of aerobic, muscular strength and muscular endurance activities and/or a dramatic change in diet,

resulting post-intervention data was excluded in the secondary performance outcomes data analysis.

Figure 5. Modified Fitnessgram Physical Activity and Diet Audit Questions

| Aerobic | Outside of the intervention with the researcher, how many of the past 7 days did you participate in any physical activity for a total of 30 to 60 minutes or over the course of a day? This includes moderate to vigorous activities (walking, slow bicycling, or outdoor play) as well as vigorous activities (jogging, active games, or active sports such as basketball, tennis, or soccer). (0, 1, 2, 3, 4, 5, 6, 7 days) |
|---|---|
| Muscular<br>strength and<br>endurance | Outside of the intervention with the researcher. how many of the past days did you exercise to strengthen or tone your muscles? This includes exercises such as push-ups, sit-ups, or weightlifting. (0, 1, 2, 3, 4, 5, 6, 7 days) |
| Diet | Have you changed your diet in the past 7 days? If so, please describe. |

Figure 5 is a modified physical activity and diet questionnaire from the Cooper Institute's Fitnessgram and Activitygram assessment manual to investigate additional activity and diet changes outside of the investigation [45].

*Participant attendance*. Participant attendance was observed by the researcher and measured as attended sessions divided by total sessions offered. Based on systematic reviews and meta-analyses [46, 47], 80% was selected as an acceptable attendance threshold.

Adverse events. Adverse events were recorded during the intervention by the participants on workout documents and by observations from the primary researcher. The primary researcher used no adverse events as an acceptable threshold.

Participant experience. Participant experience was assessed by utilizing the validated short form 4 item Physical Activity Enjoyment Scale (PACES-S) survey for adolescents [48]. Participants answered 4 items including: "I enjoyed it; I find it pleasurable; It is very pleasant; and It feels good" by responding with the five-point Likert scale ranging from 1= "strongly disagree" to 5 = "strongly agree". To further investigators' depth of understanding, participant experience was also assessed by a follow up interview concluding the intervention. Please see qualitative assumptions, interview process and qualitative data analysis section below for further details.

## **Progression criteria**

Of the above feasibility measures, selected outcomes were used as key markers to assess if further investigations were warranted for the future. The following criteria for evaluating feasibility are below:

- 1. No adverse events related to the intervention treatment.
- 2. Sample size of 30 participants per trial.
- 3. Consent rate no less than 80%.
- 4. Retention rate no less than 80%.
- 5. Attendance rates no less than 80%.

If all five criteria were met, then further investigations can continue without modification. If three to four criteria were met, then further investigations can continue with modifications. If two or less criteria were met, the study is assessed as not feasible.

## **Secondary outcomes**

All secondary outcome assessments were taken pre and post-intervention. Testing protocols required participants to avoid strenuous physical activity 48 hours prior to testing days.

Assessments took a single session to complete and all participants were tested within similar time periods.

*Bioelectric Impedance Analyzer*. In a separate private room, one participant at a time weighed themselves on a certified scale. Participants used the handheld Omron model HBF-306 to enter their weight, age, sex and activity level. Resulting BMI and body fat percentage data was recorded. Omron HBF-306 has been shown to be a reliable tool to track body composition over time [49].

Isometric lower body pull. Using the Baseline 12-0400 Back-Leg-Chest dynamometer participants stood up-right and feet hip width apart on the dynamometer platform with the chain adjusted so the handle was at the intra-articular space of the knee joint. Participants were instructed to grip the handle evenly at the center then produce a maximal 5 sec pull keeping the back from bending and arms straight. Participants were allowed to rest 30 sec between attempts. Participants had one practice attempt for familiarization purposes and then the best score of the three following attempts were recorded. Prior research has established reasonable test-retest reproducibility of the Baseline 12-0400 Back-Leg-Chest dynamometer in adolescent populations [50].

90° push-up. Participants were paired; participant 1 performed the test while participant 2 recorded the number of push-ups. Participants performed the assessment in accordance with the Cooper Institute's procedures [45]. Participant 1 assumed a prone plank position with hands slightly outside of shoulders, fingers stretched out and legs straight with a slight gap. While performing push-ups, the participants' back maintained a straight line from head to ankles. Participants started by lowering their body until the upper arms became parallel to the ground. The participant then extended their arms straight pushing their body up. This movement was

performed every three seconds by metronome and repeated until failure. Participants were allowed one form correction and two form corrections resulted in test termination. Form corrections included participants stopping to rest, a failure to maintain a straight back, achieving proper depth or fully extending the arms. Prior research notes the acceptable reliability of the push-up assessment in males and females [51].

Modified Pull-up. Participants performed the modified pull-up test in accordance with Cooper Institute's procedure [45]. Participants placed a barbell in a squat rack so that the barbell was one to two inches away from participant's reach while supine on the ground. A band was then placed seven to eight inches below the barbell. Participants started the assessment by overhand gripping the barbell and creating a straight line from head to heels so that only the heels were in ground contact. Participants then pulled their body toward the barbell until the chin was above the band. This movement was performed every three seconds by metronome and repeated until failure. Participants were allowed one form of correction and two form corrections would result in test termination. Form corrections included participants stopping to rest, failure to maintain a straight line, achieve proper depth and fully extending the arms.

PACER. To assess cardiovascular fitness, the Progressive Aerobic Cardiovascular Endurance Run (PACER) assessment was used. Prior to the start of assessment, the primary investigator measured and marked a designated 20-meter distance in the gymnasium for testing. Participants were briefed on the assessment guidelines and participated in one practice opportunity prior to the official assessment. Once familiarized, participants ran the 20-meter distance in accordance to PACER cadences from the Cooper Institute for as long as possible. The test was terminated when the participant voluntarily stopped due to fatigue or when two laps were missed. The primary researcher recorded total number of successful levels. Once

completed, the primary researcher computed predicted peak  $VO_2$  by using  $VO_2$ peak = 0.353(Laps) - 1.121(Age) + 45.619. This equation has been shown to have moderately strong linear relationships compared to measured  $VO_2$  peak of adolescents [52].

## Quantitative data analysis

Non-parametric analyses of primary and secondary outcomes were used due to the small sample size. Wilcoxon signed rank tests were used to test significance of pre and post-intervention data within treatment groups. Reports of Wilcoxon signed rank included medians, inner quartile ranges, z scores and p-values. Two sample Wilcoxon rank sum (Mann-Whitney) tests were used to test significance between treatment group differences. Reports of Wilcoxon rank-sum (Mann-Whitney) tests included medians, inner quartile ranges, U statistic and p-values. Due to an underpowered sample, effect sizes were calculated for all secondary outcome statistical tests. Given the exploratory nature of this study and the small sample, effect sizes may be more useful in guiding future research. Effect sizes were interpreted as small if r = 0.2 - 0.5, medium if r = 0.5 - 0.8 medium and large if r > 0.8. Statistical package STATA (version; BE 18.0, StataCorp, College Station, Texas, USA) was used and Alpha level was set at P < 0.05.

## **Qualitative assumptions**

Following quantitative data analysis, a constructivist paradigm was utilized for the qualitative phase. Hatch [53] depicts the ontological assumption (nature of reality) in a constructivist paradigm as "multiple realities are constructed". In a constructivist paradigm the epistemological assumption (nature of data) is that data is collected in close, personal and interactive settings. Researchers in this paradigm let the participants drive the investigation to explain their perceived reality without the addition of the researcher's influence. Thus, the

axiological assumption (value of data) is subjective and relative to the participant. These realities are important to consider as perceptions may influence how the participant behaves.

#### **Interview methods**

Participants were invited to a recorded interview for 30 min on Zoom. The interview followed a piloted semi-structured interview guide (Figure 6) created by the primary researcher to further understand participant experiences of the training protocols. Participants were given pseudonyms to protect their identity.

# Figure 6. Interview Guide

# **Background** info

Do you enjoy being active, if so why?

What about weightlifting do you find appealing?

Explain to me why you wanted to sign up for this study.

#### Participant experience

Did the timing of the workout sessions work well for you? Why or why not?

Tell me about some of the factors, if any, that made it difficult to attend.

Were there aspects of the workout sessions that you enjoyed and if so why?

Were there aspects of the workout sessions that you disliked and if so why?

In what ways did participating in this study benefit you?

In what ways did participation in this study not benefit you?

Tell me about some parts of the program, if any, that made it challenging to complete as directed.

If anything, what would you change regarding the workout sessions?

In general, how would you describe your experience participating in this study?

Figure 6 shows the semi-structured follow up interview guide.

# Qualitative data analysis

Once interviews were concluded, thematic analysis as described by Terry and colleagues [54] was conducted to analyze data. The primary researcher familiarized himself with the data by viewing recorded interviews and checking transcripts for correct transcription. Initial codes were then generated by highlighting test segments relevant to the study aims examining participant experiences. Codes were grouped into initial themes based on their underlying conceptual similarities. Themes were then reviewed and revised to generate three final themes: "It was a positive experience", "workout difficulty and duration", and "barriers". Extracts of interviews were used to support reported themes.

#### References

- Faigenbaum AD, Kraemer WJ, Blimkie CJ, Jeffreys I, Micheli LJ, Nitka M, Rowland TW. Youth resistance training: updated position statement paper from the National Strength and Conditioning Association. The Journal of Strength & Conditioning Research. 2009 Aug 1;23:S60-79.
- 2. Faigenbaum AD, Geisler S. The promise of youth resistance training. B&G Bewegungstherapie Und Gesundheitssport. 2021 Apr;37(02):47-51.
- 3. Sigal RJ, Alberga AS, Goldfield GS, Prud'homme D, Hadjiyannakis S, Gougeon R, Phillips P, Tulloch H, Malcolm J, Doucette S, Wells GA. Effects of aerobic training, resistance training, or both on percentage body fat and cardiometabolic risk markers in obese adolescents: the healthy eating aerobic and resistance training in youth randomized clinical trial. JAMA Pediatrics. 2014 Nov 1;168(11):1006-14.
- Shaibi GQ, Cruz ML, Ball GD, Weigensberg MJ, Salem GJ, Crespo NC, Goran MI.
   Effects of resistance training on insulin sensitivity in overweight Latino adolescent males.
   Medicine and science in sports and exercise. 2006 Jul 1;38(7):1208.
- 5. Naylor LH, Watts K, Sharpe JA, Jones TW, Davis EA, Thompson A, George K, Ramsay JM, O'Driscoll G, Green DJ. Resistance training and diastolic myocardial tissue velocities in obese children. Medicine and science in sports and exercise. 2008 Dec 1;40(12):2027-32.
- Moraes E, Fleck SJ, Dias MR, Simão R. Effects on strength, power, and flexibility in adolescents of nonperiodized vs. daily nonlinear periodized weight training. The Journal of Strength & Conditioning Research. 2013 Dec 1;27(12):3310-21.

- 7. Santos EJ, Janeira MA. The effects of resistance training on explosive strength indicators in adolescent basketball players. The journal of strength & conditioning research. 2012

  Oct 1;26(10):2641-7.
- 8. Sander A, Keiner M, Wirth K, Schmidtbleicher D. Influence of a 2-year strength training programme on power performance in elite youth soccer players. European journal of sport science. 2013 Sep 1;13(5):445-51.
- Keiner M, Sander A, Wirth K, Schmidtbleicher D. Long-term strength training effects on change-of-direction sprint performance. The Journal of Strength & Conditioning Research. 2014 Jan 1;28(1):223-31.
- 10. Zwolski C, Quatman-Yates C, Paterno MV. Resistance training in youth: laying the foundation for injury prevention and physical literacy. Sports health. 2017 Sep;9(5):436-43.
- 11. Lloyd RS, Faigenbaum AD, Stone MH, Oliver JL, Jeffreys I, Moody JA, Brewer C, Pierce KC, McCambridge TM, Howard R, Herrington L. Position statement on youth resistance training: the 2014 International Consensus. British journal of sports medicine. 2014 Apr 1;48(7):498-505.
- 12. Zhang X, Jiang C, Zhang X, Chi X. Muscle-strengthening exercise and positive mental health in children and adolescents: An urban survey study. Frontiers in Psychology. 2022 Aug 15;13:933877.
- 13. Harveson A, Hannon J, Brusseau T, Podlog L, Chase B, Kang KD. Acute Exercise and academic achievement in high school youth. Physical Educator. 2018;75(1):25-36.

- 14. Telama R, Yang X, Leskinen E, Kankaanpää A, Hirvensalo M, Tammelin T, Viikari JS, Raitakari OT. Tracking of physical activity from early childhood through youth into adulthood. Medicine & Science in Sports & Exercise. 2014 May 1;46(5):955-62.
- 15. Huotari P, Nupponen H, Mikkelsson L, Laakso L, Kujala U. Adolescent physical fitness and activity as predictors of adulthood activity. Journal of sports sciences. 2011 Aug 1;29(11):1135-41.
- 16. Michael SL. Dietary and Physical Activity Behaviors in 2021 and Changes from 2019 to 2021 Among High School Students—Youth Risk Behavior Survey, United States, 2021. MMWR supplements. 2023;72.
- 17. Jenkinson KA, Benson AC. Barriers to providing physical education and physical activity in Victorian state secondary schools. Australian Journal of Teacher Education (Online). 2010 Jan;35(8):1-7.
- 18. Sharp CA, McNarry MA, Eddolls WT, Koorts H, Winn CO, Mackintosh KA. Identifying facilitators and barriers for adolescents participating in a school-based HIIT intervention: the eXercise for asthma with commando Joe's®(X4ACJ) programme. BMC Public Health. 2020 Dec;20:1-1.
- 19. Aspen Institute. National Student Survey Analysis[Internet]. Resonant Education; 2022; cited 2023 Jan 8]. Available from: https://www.aspeninstitute.org/wp-content/uploads/2021/11/Aspen-National-Student-Survey-FINAL-Report.pdf
- 20. Peacock J, Finn K, Bowling A. HIIT and Resistance Training Effects on Learning-related Outcomes in Underserved School Children. Int. J. Phys. Educ. Fit. Sports. 2022;11(1):1-9.

- 21. Seo YG, Lim H, Kim Y, Ju YS, Choi YJ, Lee HJ, Jang HB, Park SI, Park KH. Effects of circuit training or a nutritional intervention on body mass index and other cardiometabolic outcomes in children and adolescents with overweight or obesity. PLoS One. 2021 Jan 28;16(1):e0245875.
- 22. Winn CO, Mackintosh KA, Eddolls WT, Stratton G, Wilson AM, McNarry MA, Davies GA. Effect of high-intensity interval training in adolescents with asthma: the eXercise for asthma with Commando Joe's®(X4ACJ) trial. Journal of Sport and Health Science. 2021 Jul 1;10(4):488-98.
- 23. Costigan SA, Eather N, Plotnikoff RC, Hillman CH, Lubans DR. High-intensity interval training for cognitive and mental health in adolescents. Med Sci Sports Exerc. 2016 Oct 1;48(10):1985-93.
- 24. Mezcua-Hidalgo A, Ruiz-Ariza A, Suárez-Manzano S, Martínez-López EJ. 48-hour effects of monitored cooperative high-intensity interval training on adolescent cognitive functioning. Perceptual and motor skills. 2019 Apr;126(2):202-22
- 25. Paoli A, Pacelli F, Bargossi AM, Marcolin G, Guzzinati S, Neri M, Bianco A, Palma A. Effects of three distinct protocols of fitness training on body composition, strength and blood lactate. J Sports Med Phys Fitness. 2010 Mar 1;50(1):43-51.
- 26. Brown, LE & National Strength & Conditioning Association. Strength Training. 2nd ed. Champaign (IL): Human Kinetics; 2017.
- 27. Faigenbaum AD, Ratamess NA, McFarland J, Kaczmarek J, Coraggio MJ, Kang J, Hoffman JR. Effect of rest interval length on bench press performance in boys, teens, and men. Pediatric exercise science. 2008 Nov 1;20(4):457-69.

- 28. Channell BT, Barfield JP. Effect of Olympic and traditional resistance training on vertical jump improvement in high school boys. The Journal of Strength & Conditioning Research. 2008 Sep 1;22(5):1522-7.
- 29. Alcaraz PE, Sánchez-Lorente J, Blazevich AJ. Physical performance and cardiovascular responses to an acute bout of heavy resistance circuit training versus traditional strength training. The Journal of Strength & Conditioning Research. 2008 May 1;22(3):667-71.
- 30. Thompson BJ, Stock MS, Mota JA, Drusch AS, DeFranco RN, Cook TR, Hamm MA. Adaptations associated with an after-school strength and conditioning program in middle-school-aged boys: A quasi-experimental design. The Journal of Strength & Conditioning Research. 2017 Oct 1;31(10):2840-51.
- 31. Kretschmann R. Effects of an 8-week after-school resistance program in secondary school students. Journal of Physical Education and Sport. 2023 Jun 1;23(6):1376-84.
- 32. Alcaraz PE, Perez-Gomez J, Chavarrias M, Blazevich AJ. Similarity in adaptations to high-resistance circuit vs. traditional strength training in resistance-trained men. The Journal of Strength & Conditioning Research. 2011 Sep 1;25(9):2519-27.
- 33. Paoli A, Moro T, Marcolin G, Neri M, Bianco A, Palma A, Grimaldi K. High-Intensity Interval Resistance Training (HIRT) influences resting energy expenditure and respiratory ratio in non-dieting individuals. Journal of translational medicine. 2012

  Dec;10:1-8.
- 34. Ramos-Campo DJ, Rubio-Arias JÁ, Freitas TT, Camacho A, Jiménez-Diaz JF, Alcaraz PE. Acute physiological and performance responses to high-intensity resistance circuit training in hypoxic and normoxic conditions. The Journal of Strength & Conditioning Research. 2017 Apr 1;31(4):1040-7.

- 35. Marín-Pagán C, Blazevich AJ, Chung LH, Romero-Arenas S, Freitas TT, Alcaraz PE. Acute physiological responses to high-intensity resistance circuit training vs. traditional strength training in soccer players. Biology. 2020 Nov 7;9(11):383.
- 36. Freitas TT, Calleja-González J, Alarcón F, Alcaraz PE. Acute effects of two different resistance circuit training protocols on performance and perceived exertion in semiprofessional basketball players. The Journal of Strength & Conditioning Research. 2016 Feb 1;30(2):407-14.
- 37. Romero Arenas S, Blazevich AJ, Martínez Pascual M, Pérez Gómez J, Luque AJ, López Román FJ, Alcaraz Ramón PE. Effects of high-resistance circuit training in an elderly population. Experimental Gerontology. 2013;48(3).
- 38. El-Kotob R, Giangregorio LM. Pilot and feasibility studies in exercise, physical activity, or rehabilitation research. Pilot and feasibility studies. 2018 Dec;4:1-7.
- 39. Helms ER, Byrnes RK, Cooke DM, Haischer MH, Carzoli JP, Johnson TK, Cross MR, Cronin JB, Storey AG, Zourdos MC. RPE vs. percentage 1RM loading in periodized programs matched for sets and repetitions. Frontiers in physiology. 2018 Mar 21;9:247.
- 40. Shattock K, Tee JC. Autoregulation in resistance training: a comparison of subjective versus objective methods. The Journal of Strength & Conditioning Research. 2022 Mar 1;36(3):641-8.
- 41. Pfledderer CD, von Klinggraeff L, Burkart S, da Silva Bandeira A, Lubans DR, Jago R, Okely AD, van Sluijs EM, Ioannidis JP, Thrasher JF, Li X. Consolidated guidance for behavioral intervention pilot and feasibility studies. Pilot and Feasibility Studies. 2024 Apr 6;10(1):57.

- 42. Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharmaceutical Statistics: The Journal of Applied Statistics in the Pharmaceutical Industry. 2005

  Oct;4(4):287-91.
- 43. Jacques RM, Ahmed R, Harper J, Ranjan A, Saeed I, Simpson RM, Walters SJ.

  Recruitment, consent and retention of participants in randomised controlled trials: a review of trials published in the National Institute for Health Research (NIHR) Journals Library (1997–2020). BMJ open. 2022 Feb 1;12(2):e059230.
- 44. Schulz KF, Grimes DA. Sample size slippages in randomised trials: exclusions and the lost and wayward. The Lancet 2002 Mar 02;359(9308):781-785.
- 45. Welk G, Meredith MD. Fitnessgram and Activitygram Test Administration Manual. 4th ed. Champian (IL): Human Kinetics; 2010.
- 46. Weston KS, Wisloff U, Coombes JS. High-intensity interval training in patients with lifestyle-induced cardiometabolic disease: a systematic review and meta-analysis. Br J Sports Med. 2014;48:1227–34. https://doi.org/10.1136/bjsports-2013-092576.
- 47. De Nardi AT, Tolves T, Lenzi TL, Signori LU, da Silva AM. High-intensity interval training versus continuous training on physiological and metabolic variables in prediabetes and type 2 diabetes: a meta-analysis. Diabetes research and clinical practice. 2018 Mar 1;137:149-59.
- 48. Chen C, Weyland S, Fritsch J, Woll A, Niessner C, Burchartz A, Schmidt SC, Jekauc D. A short version of the physical activity enjoyment scale: development and psychometric properties. International Journal of Environmental Research and Public Health. 2021 Oct 20;18(21):11035.

- 49. Fahs CA, Boring J, LeVault L, Varner W, Beck M. The accuracy of commercially available upper and lower body bioelectrical impedance analyzers in men and women. Biomedical Physics & Engineering Express. 2020 Apr 22;6(3):035017.
- 50. Ten Hoor GA, Musch K, Meijer K, Plasqui G. Test-retest reproducibility and validity of the back-leg-chest strength measurements. Isokinetics and Exercise Science. 2016 Jan 1;24(3):209-16.
- 51. Hashim A, Madon MS. Objectivity, reliability and validity of the 90° push-ups test protocol among male and female students of sports science program. International Journal of Sport and Health Sciences. 2012 Jun 23;6(6):1068-71.
- 52. Burns RD, Hannon JC, Brusseau TA, Eisenman PA, Saint-Maurice PF, Welk GJ, Mahar MT. Cross-validation of aerobic capacity prediction models in adolescents. Pediatric exercise science. 2015 Aug 1;27(3):404-11.
- 53. Hatch, JA. Doing qualitative research in education settings. Albany (NY): State
  University of New York; 2002. Chapter 1, Deciding to do a Qualitative Study; p. 1-36.
- 54. Terry G, Hayfield N, Clarke V, Braun V. Thematic analysis. The SAGE handbook of qualitative research in psychology. 2017 Jun 30;2(17-37):25.
- 55. Zhao M, Liu S, Han X, Li Z, Liu B, Chen J, Li X. School-Based Comprehensive Strength Training Interventions to Improve Muscular Fitness and Perceived Physical Competence in Chinese Male Adolescents. BioMed Research International. 2022;2022(1):7464815.
- 56. Garst BA, Bowers EP, Stephens LE. A randomized study of CrossFit Kids for fostering fitness and academic outcomes in middle school students. Evaluation and program planning. 2020 Dec 1;83:101856.

- 57. 1991–2023 High School Youth Risk Behavior Survey Data. Centers for Disease Control and Prevention. 2024. http://yrbs-explorer.services.cdc.gov/. Accessed 1 Oct 2024.
- 58. Campbell IG, Burright CS, Kraus AM, Grimm KJ, Feinberg I. Daytime sleepiness increases with age in early adolescence: a sleep restriction dose–response study. Sleep. 2017 May 1;40(5):zsx046.
- 59. Baum KT, Desai A, Field J, Miller LE, Rausch J, Beebe DW. Sleep restriction worsens mood and emotion regulation in adolescents. Journal of Child Psychology and Psychiatry. 2014 Feb;55(2):180-90
- 60. Jiang F, VanDyke RD, Zhang J, Li F, Gozal D, Shen X. Effect of chronic sleep restriction on sleepiness and working memory in adolescents and young adults. Journal of Clinical and Experimental Neuropsychology. 2011 Oct 1;33(8):892-900.
- 61. Mitchell JA, Rodriguez D, Schmitz KH, Audrain-McGovern J. Sleep duration and adolescent obesity. Pediatrics. 2013 May 1;131(5):e1428-34.
- 62. Santiago LC, Lyra MJ, Germano-Soares AH, Lins-Filho OL, Queiroz DR, Prazeres TM, Mello MT, Pedrosa RP, Falcão AP, Santos MA. Effects of strength training on sleep parameters of adolescents: a randomized controlled trial. The Journal of Strength & Conditioning Research. 2022 May 1;36(5):1222-7.